CLINICAL TRIAL: NCT05103449
Title: Effect of Video-Based Coaching on Resident Laparoscopic Surgical Skills: A Randomized Controlled Trial
Brief Title: Effect of Video-Based Coaching on Resident Laparoscopic Surgical Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Lisa Chao, Assistant Professor, Department of Obstetrics and Gynecology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STU-2021-0805
Record Dates: First submitted 2021-10-01; First posted 2021-11-02 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Laparoscopic Salpingectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Attending physicians evaluating the laparoscopic salpingectomy videos will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Video Coaching) (No Intervention): Control Group (No Video Coaching)
- Experimental Group (Video Coaching) (Experimental): Video-based coaching group
  Interventions: Other: Video Coaching

INTERVENTIONS:
Other: Video Coaching — Video-based coaching sessions after salpingectomy 1 and 2
  Arms: Experimental Group (Video Coaching)

SUMMARY:
Randomized controlled trial to evaluate the effect of video-based coaching on Obstetrics and Gynecology residents' efficiency, proficiency, and confidence in performing laparoscopic salpingectomy.

DETAILED DESCRIPTION:
University of Texas Southwestern PGY-1 and PGY-2 Obstetrics and Gynecology residents will be scheduled to complete a 4-week gynecology rotation at Parkland Memorial Hospital. After completing the pre-survey, trainees will be randomized into either the control or experimental group (video coached group) stratified by PGY (Post-Graduate Year) level. Minimum group sample sizes of 9 and 9 to achieve 90% power to detect a difference of 5.0 in a design with 3 repeated measurements having a Simple covariance structure when the standard deviation is 5.4 and the alpha level is 0.05. The control group will be video recorded performing three laparoscopic salpingectomy procedures as scheduled during the 4-week block. The control group will not participate in video coaching sessions. The experimental group will be video recorded performing three laparoscopic salpingectomy procedures as scheduled during the block. After the first and second laparoscopic salpingectomy, the experimental group of residents will review their video recording and receive a video coaching session by a minimally invasive gynecologic surgery (MIGS) attending physician prior to the next surgery. All three video recordings for each participant (control and experimental group) will be graded using Global Operative Assessment of Laparoscopic Skills (GOALS) and Objective Structured Assessment of Laparoscopic Salpingectomy (OSA-LS) criteria by two attending physicians not involved in the surgeries or coaching. Each surgery will be blinded to the group allocation and the week definition. Participants will not be given the assessment score and the score will not affect evaluations. After the third laparoscopic salpingectomy, trainees will fill out a post-course survey to determine if the video-based coaching course improved their proficiency and confidence in laparoscopic gynecologic surgery. They will also watch their own laparoscopic salpingectomy video recording and self-grade their skills using the GOALS and OSA-LS criteria that will be provided in the post-survey.

ELIGIBILITY:
Inclusion Criteria:

* PGY-1 and PGY-2 UTSW OB/GYN Residents during their Gynecology Block

Exclusion Criteria:

* Residents who have previously participated in the study
* PGY-3 or PGY-4 residents

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
GOALS scores on participants' last salpingectomy video | From Week 1 to Week 4
  Global Operative Assessment of Laparoscopic Skills (GOALS) is a validated assessment scale for laparoscopic surgery. GOALS has maximum of 5 points in each of 5 categories, highest score = 25.
OSA-LS scores on participants' last salpingectomy video | From Week 1 to Week 4
  Objective Structured Assessment of Laparoscopic Salpingectomy (OSA-LS) is a validated assessment scale for laparoscopic salpingectomy. OSA-LS has maximum of 5 points in each of 10 categories, highest score = 50.

SECONDARY OUTCOMES:
Time to complete salpingectomy | From Week 1 to Week 4
  Time to complete salpingectomy from start of procedure (instruments inserted to begin salpingectomy) to end of procedure (removal of fallopian tube from trocar)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Chao, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muir TM, Pruszynski J, Kho KA, Ramirez CI, Donnellan NM, Chao L. Video-Based Coaching for Laparoscopic Salpingectomy: A Randomized Controlled Trial. Obstet Gynecol. 2024 Sep 1;144(3):358-365. doi: 10.1097/AOG.0000000000005677. Epub 2024 Jul 25. PMID 39053009